CLINICAL TRIAL: NCT05228977
Title: Prevalence of Cervical Extension of the Thymus in Children- A Prospective Study
Brief Title: Prevalence of Cervical Extension of the Thymus in Children
Acronym: CET
Status: Completed | Type: Observational
Sponsor: Kabul University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Habib Ahmad Esmat, Research committee, Kabul University of Medical Sciences
Other Study IDs: 0002
Record Dates: First submitted 2022-01-26; First posted 2022-02-08 (Actual); Last update posted 2022-02-08 (Actual); Status verified 2022-02

CONDITIONS: Prevalence of Cervical Extension of the Thymus
Keywords: Thymus; Cervical extension; Pediatrics;

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This prospective, observational study included all pediatric patients who were referred to the radiology department for neck ultrasonography between August-October 2018. A high-frequency probe was implemented and 220 patients were examined.

DETAILED DESCRIPTION:
This prospective single-centered study was approved by the Institutional Review Board for Ethical Issues in Clinical Research and is compatible with the Declaration of Helsinki. The patients referred to the radiology department for the neck US with various clinical indications between August-October 2018 were included in the study. The informed consent was taken from the parents of the patients. The patients who had any systemic illness, were treated for malignancy or had any history of lower neck or chest surgery, were excluded.

The neck US was performed by two radiologists. The length of the extended thymus, from the upper margin of the manubrium to the superior edge of the thymic tissue on the transverse plane, was measured in millimeters and recorded.

al analysis of the data was performed in SPSS, Version 24 program (IBM, Armonk, New York). Pearson Chi-Square Test was used in comparing categorical data between groups.

ELIGIBILITY:
Inclusion Criteria:

* The patients referred to the radiology department for the neck US with various clinical indications between August-October 2018 were included in the study.

Exclusion Criteria:

* The patients who had any systemic illness, were treated for malignancy, or had any history of lower neck or chest surgery, were excluded.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients referred to the radiology department for the neck US with various clinical indications between August-October 2018 were included in the study.
Sampling Method: Non-Probability Sample
Enrollment: 220 (Actual)
Dates: Start 2018-08-01 (Actual); Primary Completion 2018-10-01 (Actual); Study Completion 2018-10-30 (Actual)

PRIMARY OUTCOMES:
0 | 3 months
  As our trial has no intervention, so there were no positive or negative primary effects

CONTACTS AND LOCATIONS:
Overall Officials: Mohammad wali Nasary, MD, Study Director — KMUs
Locations (2):
- Afghanistan (2):
  - Habib Ahmad Esmat, Kabul, None Selected
  - KUMs, Kabul